CLINICAL TRIAL: NCT01637532
Title: Chemo-Immunotherapy: Observational Trial of Carboplatin-pegylated Liposomal Doxorubicin (PLD) or Doxorubicin Combination Chemotherapy With Tocilizumab, a Humanized Monoclonal Antibody Against the Human Interleukin-6 (IL-6) Receptor, and Pegylated Interferon Alpha (Peg-Intron) for Patients With Recurrent Ovarian Cancer.
Brief Title: Feasibility of the Combination of Chemotherapy (Carbo/Caelyx or Carbo/Doxorubicin) With Tocilizumab (mAb IL-6R) and Peg-Intron in Patients With Recurrent Ovarian Cancer
Acronym: PITCH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, J.R. Kroep, MD, PhD, Leiden University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PITCH trial
Record Dates: First submitted 2012-04-15; First posted 2012-07-11 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Recurrent Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — tocilizumab; Carboplatin; liposomal doxorubicin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Other): Carboplatin/Caelyx
  Interventions: Drug: Carboplatin and Caelyx or doxorubicin
- Group 2 (Experimental): Carboplatin/Caelyx or doxorubicin plus Tocilizumab
  Interventions: Drug: tocilizumab and interferon alpha 2-b; Drug: Carboplatin and Caelyx or doxorubicin
- Group 3 (Experimental): Carboplatin/Caelyx or doxorubicin plus Tocilizumab plus Peg-Intron
  Interventions: Drug: tocilizumab and interferon alpha 2-b; Drug: Carboplatin and Caelyx or doxorubicin

INTERVENTIONS:
Drug: tocilizumab and interferon alpha 2-b — During first three chemotherapy cycles, tocilizumab and/or Peg-Intron are added.
  Tocilizumab is given in a dose-escalation scheme (1,2,4,8mg/kg n=3) and Peg-Intron is adminstered subcutaneously 1.0ug/kg
  Arms: Group 2; Group 3
Drug: Carboplatin and Caelyx or doxorubicin — Standard chemotherapeutic care given in every arm as standard care. A total of 6 cycles is the aim.

SUMMARY:
The purpose of this interventional study is to determine the feasibility to combine standard chemotherapy (Carbo/Caelyx or doxorubicin) for recurrent ovarian cancer with immunotherapy (Tocilizumab and Peg-Intron).

This study combines standard chemotherapy Carboplatin-Caelyx or doxorubicin with a monoclonal antibody against IL-6R (tocilizumab). High IL-6 levels correlate with poor prognosis and chemoresistance in ovarian cancer patients. In cases of chemoresistant ovarian cancer, therefore, modulation of the IL-6 pathway, by blocking the IL-6 receptor, may represent a promising strategy to both abolish drug resistance and amplify host immunity in patients with recurrent ovarian cancer. Blockade of the IL-6/IL-6R pathway may enhance immunogenic cell death and restore local normal DC maturation. In addition, the use of interferon-alpha (Peg-Intron) allows the full maturation of DC, thereby enhancing the anti-tumor response.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven epithelial ovarian cancer
* Progression of disease or relapse after previous therapy with platinum
* Measurable disease (RECIST 1.1) or elevated CA125 > 2 times the upper normal limit (UNL) within 3 months and confirmed
* Age ≥18 years
* WHO performance status 0-2
* Adequate bone marrow function: WBC ≥3.0 x 109/l, neutrophils ≥1.5 x 109/l, platelets ≥100 x 109/l
* Adequate liver function: bilirubin ≤1.5 x UNL range, ALAT and/or ASAT

  * 2.5 x UNL (<5x UNL in case of liver metastases), Alkaline Phosphatase ≤5 x UNL
* Adequate renal function: the calculated creatinine clearance should be

  * 50 mL/min
* Survival expectation > 3 months
* Patients must be accessible for treatment and follow-up
* Written informed consent according to the local Ethics Committee requirements

Exclusion Criteria:

* Chemotherapy within past 3 months
* Previous malignancy within 5 years, with exception of a history of a previous basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix
* Serious other diseases as recent myocardial infarction, clinical signs of cardiac failure or clinically significant arrhythmias
* Known hypersensitivity reaction to any of the components of the treatment
* Pregnancy or lactating
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent
* Infection with tuberculosis and hepatitis B or C

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The feasibility (NCI-CTCv4.0) to combine carboplatin and PLD or doxorubicin with tocilizumab as well as with tocilizumab and Peg-Intron | two years
  The safety (NCI-CTCv4.0)and efficacy (immune-monitoring)of the new combination will be measured .

SECONDARY OUTCOMES:
The effect of chemo-immunotherapy on the immune system | two years
  Study the effect of chemo-immunotherapy on the immune system by assessing changes in plasma signature (eg IL6, IL8, VEGF, CRP) dendritic cell phenotype and T- and B-cell responses to known tumor antigens in ovarian cancer (eg NY-ESO, p53), antibodies to antigens associated with immunogenic cell death (CRT, HMGB1) and in tumor tissue by gene array
The relation between anti-tumor immunity and clinical outcome | two years
  Study the relation between anti-tumor immunity and clinical outcome (response (RECIST 1.1), progression free survival (PFS) and overall survival(OS))

CONTACTS AND LOCATIONS:
Overall Officials: G Blecourt, Study Director — LUMC
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Derived] Dijkgraaf EM, Santegoets SJ, Reyners AK, Goedemans R, Wouters MC, Kenter GG, van Erkel AR, van Poelgeest MI, Nijman HW, van der Hoeven JJ, Welters MJ, van der Burg SH, Kroep JR. A phase I trial combining carboplatin/doxorubicin with tocilizumab, an anti-IL-6R monoclonal antibody, and interferon-alpha2b in patients with recurrent epithelial ovarian cancer. Ann Oncol. 2015 Oct;26(10):2141-9. doi: 10.1093/annonc/mdv309. Epub 2015 Jul 27. PMID 26216383